CLINICAL TRIAL: NCT03543761
Title: Evaluation of Low-intensity Shockwave Therapy for Non-bacterial Prostatitis/Pelvic Pain Syndrome: a Triple-blind Randomized Controlled Trial
Brief Title: Low-intensity Shockwave Therapy for Non-bacterial Prostatitis/Pelvic Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for the Study of Urological Diseases, Greece (Other)
Responsible Party: Principal Investigator, Dimitrios Hatzichristou, President, Institute for the Study of Urological Diseases Theesaloniki, Greece, Institute for the Study of Urological Diseases, Greece
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1340/2018
Record Dates: First submitted 2018-04-25; First posted 2018-06-01 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Chronic Prostatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Sham Comparator): Sham group
  Interventions: Device: Dornier Aries 2 device
- B (Active Comparator): LiST active treatment group
  Interventions: Device: Dornier Aries 2 device
- C (Active Comparator): LiST active treatment group
  Interventions: Device: Dornier Aries 2 device

INTERVENTIONS:
Device: Dornier Aries 2 device — • Sham group: 6 sessions with placebo LiST probe, 1 session per week. A specific probe design, identical to the active one will allow the double blind fashion of the study.
  Arms: A
Device: Dornier Aries 2 device — LiST groups: 6 sessions with active LiS probe, 1 session per week. The ARIES 2 device by Dornier will be used with a treatment protocol: 5000 SW, energy flux density = 0.096 mJ/mm2 (energy level 7)
  Arms: B
Device: Dornier Aries 2 device — LiST groups: 6 sessions with active LiS probe, 1 session per week. The ARIES 2 device by Dornier will be used with a treatment protocol: 5000 SW, energy flux density = 0.096 mJ/mm2 (energy level 7)
  Arms: C

SUMMARY:
The aim of the study is to investigate and compare the treatment efficacy and safety of ESWT vs sham treatment for CP/CPPS patients.This is a triple-blind, randomized, parallel group sham-controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must 18 to 60 years of age.
2. Participant has signed and dated the appropriate Informed Consent document.
3. Participant has had a clinical diagnosis of CP/CPPS defined as symptoms of discomfort or pain in the perineal or pelvic region for at least a three (3) month period within the last six (6) months

Exclusion Criteria:

1. Participant has evidence of facultative Gram negative or enterococcus with a value of ≥ 1000 CFU/ml in mid-stream urine (VB2).
2. Participant has a history of prostate, bladder or urethral cancer.
3. Participant has undergone pelvic radiation or systemic chemotherapy.
4. Participant has undergone intravesical chemotherapy.
5. Participant has unilateral orchialgia without pelvic symptoms, active urethral stricture or bladder stones, or any other urological condition associated with LUTS, any neurological disease or disorder affecting the bladder.
6. Participant has undergone prostate surgery or treatment.
7. Participant with penile or urinary sphincter implants.
8. Participant has been diagnosed with cancer during the last 5 years, or had any surgery in the pelvis.
9. Participant has a neurological impairment or psychiatric disorder preventing his understanding of consent and his ability to comply with the protocol.
10. PI-RADS score 4-5 in the baseline prostate mpMRI
11. PI-RADS score 3, PSA>3 and age > 40 years
12. Positive (suspicious for malignancy) DRE.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
The difference between the LiST and sham group in the change of the pain domain of NIH-CPSI score | from baseline to 12 weeks after final treatment.
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special pain domain (items 1-4) and the score for this domain ranges from 0 to 21.

SECONDARY OUTCOMES:
The difference between the LiST and sham group in the change of total NIH-CPSI score (Q1-9) | baseline, 4 and 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).
The difference between the LiST and sham group in the change of urinary symptoms (Q 5-6) and quality of life domains (Q 7-9) of the NIH-CPSI score | from baseline to 4 and 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special urinary symptom domain (items 5-6) and the score for this domain ranges from 0 to 10.
The difference between the LiST and sham group in the change of quality of life domains (Q 7-9) of the NIH-CPSI score | from baseline to 4 and 12 weeks after final treatment
  CP/CPPS-related complaints will be assessed by the the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI). The questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain (items 1-4), urinary symptoms (items 5-6), and quality of life (items 7-9).Total score ranges from 0 to 35 (higher values represent worse outcome).The index provides a special quality of life domain (items 7-9) and the score for this domain ranges from 0 to 12.
The difference between the LiST and sham group in the change of IIEF-ED score | from baseline to 4 weeks after final treatment.
  It will be assessed by International Index of Erectile Function -Erectile Domain (IEF-ED) score. A questionnaire designed to evaluate erectile capabilities. The questionnaire provides a score between 5 and 30.The severity categories are: 1-10 severe ED, 10-16 moderate ED, 17-21 moderate to mild ED, 22-25 mild ED, 26-30 no ED
The difference between the LiST and sham group in the change of IPSS | from baseline to 4 weeks after final treatment.
  They will be assessed by the International Prostate Symptom Score (IPSS). A questionnaire designed to provide information on lower urinary tract symptoms and their impact on quality of life. Scores range from 0 to 35. The severity categories are: 1-7 mild, 8-19 moderate, 20-35 severe
The difference between the LiST and sham group in the change of Maximum urinary flow rate (Qmax)/ Post Void Residual (PVR) | from baseline to 4 weeks after final treatment.
  Qmax will be measured by uroflowmetry/ PVR will be measured by ultrasound
The difference between the LiST and sham group in the change of UPPOINTS phenotype- number of positive domains | from baseline to 4 weeks after final treatment.
The difference between the LiST and sham group in the the Pain Visual Analogue Scale (VAS) | at week 3, 4, 5, 6, 7 and 8
  It will be assessed by the pain VAS, right after each LIST session. Pain VAS is a unidimensional measure of pain intensity . It is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]. To avoid clustering of scores around a preferred numeric value, numbers or verbal descriptors at intermediate points are not recommended. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm)
Changes in mpMRI of the prostate | baseline and 12 weeks after treatment
Adverse events rate in all patients | 18 weeks
  Potential treatment related adverse events after the first LIST session and during the 3 month follow up period will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Hatzichristou, Prof., Principal Investigator — Institute for the Study of Urological Diseases, Thessaloniki, Greece
Locations (1):
- G.Gennimatas Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimmermann R, Cumpanas A, Miclea F, Janetschek G. Extracorporeal shock wave therapy for the treatment of chronic pelvic pain syndrome in males: a randomised, double-blind, placebo-controlled study. Eur Urol. 2009 Sep;56(3):418-24. doi: 10.1016/j.eururo.2009.03.043. Epub 2009 Mar 25. PMID 19372000
- [Background] Al Edwan GM, Muheilan MM, Atta ON. Long term efficacy of extracorporeal shock wave therapy [ESWT] for treatment of refractory chronic abacterial prostatitis. Ann Med Surg (Lond). 2017 Jan 6;14:12-17. doi: 10.1016/j.amsu.2016.12.051. eCollection 2017 Feb. PMID 28119778